CLINICAL TRIAL: NCT04418349
Title: Evaluation of Posterior Component Separation Modified TAR Technique "Transversus Abdominids Release" in the Treatment of Parastomal Hernia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R.19.07.563 - 2019/07/15
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Last update posted 2020-06-18 (Actual); Status verified 2020-05

CONDITIONS: TAR Technique

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: posterior component separation modified TAR technique "Transversus Abdominids Release" — Evaluation of posterior component separation modified TAR technique "Transversus Abdominids Release" in the treatment of parastomal hernia

SUMMARY:
Aim of the work In this study, we will evaluate posterior Evaluation of posterior component separation modified TAR technique "Transversus Abdominids Release" in the treatment of parastomal hernia. The primary outcome will be recurrence while the secondary outcome will be infection, postoperative complications (bleeding and dehiscence), pain score, operative time, hospitalization, need for drain, time for drain removal and pulmonary function test before and after surgery

ELIGIBILITY:
Inclusion Criteria:

* Adult patient fit for general anesthesia with parastomal herniation.

Exclusion Criteria:

* Patients who are unfit for general anaesthesia.
* Poor pulmonary function tests.
* Pregnant females.
* Patient younger than 18 years.
* Immunodeficiency.
* Patient with psychiatric disease disabling surgical intervention.

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-02 (Estimated)

PRIMARY OUTCOMES:
Recurrence rate | one year
  Recurrence rate of parastomal hernias

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University, Al Mansurah, Dakahlia Governorate, Egypt